CLINICAL TRIAL: NCT03782220
Title: Effects of Kinesio Taping in Patients With Somatosensory Tinnitus: A Randomized Controlled Trial
Brief Title: Effects of Kinesio Taping in Patients With Somatosensory Tinnitus
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hitit University (Other)
Responsible Party: Principal Investigator, Tuğba Atan, Assoc. Prof., Hitit University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2018-12
Record Dates: First submitted 2018-12-17; First posted 2018-12-20 (Actual); Last update posted 2018-12-20 (Actual); Status verified 2018-12

CONDITIONS: Tinnitus, Subjective
Keywords: somatosensory tinnitus; neck pain; kinesio taping
MeSH Terms: conditions — Tinnitus; Neck Pain | interventions — Athletic Tape

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Kinesio taping group (Experimental): Kinesio taping group
  * Application of kinesio taping to sternocleidomastoid, upper trapezium, levator scapulae muscles.
  * Once a week , for 4 weeks
  Interventions: Other: Kinesio tape
- Shame taping group (Placebo Comparator): Shame taping group
  * Application of kinesio band to same muscles except for the defined method which is considered to be ineffective.
  * Once a week , for 4 weeks
  Interventions: Other: Shame tape

INTERVENTIONS:
Other: Kinesio tape — The Kinesio taping ( Kinesio Tex Gold, 2in x103.3 ft) was applied to sternocleidomastoid, upper trapezium and levator scapulae muscles by the muscle inhibition technique ( from insertion to origin of a muscle) for experimental group.
  Arms: Kinesio taping group
Other: Shame tape — For the Shame taping group, a placebo taping method considered to be ineffective ( not from insertion to origin of muscles) with the same material without tension and with the neck in neutral position was used.
  Arms: Shame taping group

SUMMARY:
There is no specific treatment that can cure somatosensory tinnitus and usually conservative physical therapy modalities are used in the literature. The aim of the study is to investigate the effect of kinesio taping applied to sternocleidomastoid, upper trapezium and levator scapulae muscles on the somatosensory tinnitus associated with neck complaints.

DETAILED DESCRIPTION:
The study was designed as a prospective, randomized controlled and double blind trial.

Patients complaining of tinnitus were firstly subjected to otologic and audiologic evaluation by an otolaryngologist. Tinnitus characteristics, such as severity (Tinnitus handicap Index, tinnitus Visual Analog Scale- tinnitus VAS) , type (pulsatile/non-pulsatile), localization (unilateral/ bilateral) and the frequency (number of days with symptoms) were recorded. Patients were excluded if they had objective tinnitus, subjective tinnitus with hearing loss or Meniere's disease, vertigo, middle ear pathologies, intracranial pathologies, whiplash injury, previous cervical spinal surgery, pregnancy, infection, malignancy and if they received cervical physical rehabilitation program in the past 3 months.

Patients who diagnosed with somatosensory tinnitus and concomitant neck complaints (cervical-VAS score >2) at least 6 weeks were referred to physical medicine and rehabilitation outpatient clinic. Before the treatment, participants' demographics data including age, gender, Body-Mass Index (BMI) and cervical pain VAS score were recorded and physical examinations (cervical joint range of motion (cervical-ROM), cervical manual muscle testing (cervical-MMT) and myofascial trigger points for sternocleidomastoid, upper trapezium and levator scapulae muscles) were performed by one investigator.

Banding application performed for both groups once a week for four weeks. Tinnitus handicap index score, tinnitus VAS, ROM of the cervical joint, cervical MMT, cervical pain VAS, Neck Disability index score and myofascial trigger points of sternocleidomastoid, upper trapezium, levator scapula was evaluated in all subjects by the same investigator.

ELIGIBILITY:
Inclusion Criteria:

* Subject has somatosensory tinnitus
* Subject has concomitant neck complaints (cervical-VAS score >2) at least 6 weeks
* Subject were referred to physical medicine and rehabilitation outpatient clinic

Exclusion Criteria:

* History of objective tinnitus
* History of subjective tinnitus with hearing loss
* History of Meniere's disease
* History of vertigo
* Hiistory of middle ear pathologies
* History of intracranial pathologies
* History of whiplash injury
* History of previous cervical spinal surgery
* History of infection or malignancy
* Pregnancy
* History of having received cervical physical rehabilitation program in the past 3 months

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2017-09-20 (Actual); Primary Completion 2018-04-18 (Actual); Study Completion 2018-09-07 (Actual)

PRIMARY OUTCOMES:
Tinnitus handicap Index (THI) | 4 weeks
  The questionnaire comprises 25 items with a functional subscale (11 items), emotional subscale (9 items), and catastrophic subscale (5 items). Each question is rated as 0 (none), 2 (sometimes), or 4 (always). Total score range from 0 to 100, with higher scores indicating higher levels of perceived tinnitus handicap.
Tinnitus severity (tinnitus-VAS) | 4 weeks
  The loudness of tinnitus was graded with a10 cm of visual analog scale (VAS, 0-10 cm; 0 means no tinnitus, 10 means extremely loud tinnitus)
Cervical pain (cervical-VAS) | 4 weeks
  Pain intensity was measured with VAS which is used to measure musculoskeletal pain with very good reliability and validity (VAS, 0-10 cm; 0 means no pain, 10 means severe pain).
Neck Disability index score (NDI) | 4 weeks
  The NDI is designed to assess self - reported neck functional status. The questionnaire comprises 10 items related to pain, activities of daily living, lifting, reading, headaches, concentration, work status, driving, sleeping and recreation, each rated on a 6-point Likert scale with a final score range of 0 (no disability) to 50 (major disability). Higher scores represent greater disability

CONTACTS AND LOCATIONS:
Locations (1):
- Tuğba Atan, Çorum, Turkey (Türkiye)

REFERENCES:
- [Result] Ralli M, Altissimi G, Turchetta R, Mazzei F, Salviati M, Cianfrone F, Orlando MP, Testugini V, Cianfrone G. Somatosensory Tinnitus: Correlation between Cranio-Cervico-Mandibular Disorder History and Somatic Modulation. Audiol Neurootol. 2016;21(6):372-382. doi: 10.1159/000452472. Epub 2017 Jan 19. PMID 28099967
- [Result] Vanneste S, Plazier M, Van de Heyning P, De Ridder D. Transcutaneous electrical nerve stimulation (TENS) of upper cervical nerve (C2) for the treatment of somatic tinnitus. Exp Brain Res. 2010 Jul;204(2):283-7. doi: 10.1007/s00221-010-2304-5. Epub 2010 May 28. PMID 20505927
- [Result] Rocha CB, Sanchez TG. Efficacy of myofascial trigger point deactivation for tinnitus control. Braz J Otorhinolaryngol. 2012 Dec;78(6):21-6. doi: 10.5935/1808-8694.20120028. PMID 23306563
- [Result] Michiels S, Van de Heyning P, Truijen S, Hallemans A, De Hertogh W. Does multi-modal cervical physical therapy improve tinnitus in patients with cervicogenic somatic tinnitus? Man Ther. 2016 Dec;26:125-131. doi: 10.1016/j.math.2016.08.005. Epub 2016 Aug 26. PMID 27592038